CLINICAL TRIAL: NCT01648907
Title: French Cohort on Outcome of Recent Undifferentiated Spondyloarthritis
Brief Title: French Cohort of Undifferentiated Spondyloarthritis
Acronym: DESIR
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P070302; IDRCB 2007-A00608-45 (Other: ANSM)
Record Dates: First submitted 2012-07-20; First posted 2012-07-24 (Estimated); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: EARLY UNDIFFERENTIATED SPONDYLARTHROPATHIES
Keywords: DESIR; SPONDYLARTHRITIS; EARLY INFLAMMATORY RACHIIALGIA; BACK PAIN
MeSH Terms: conditions — Spondylarthritis; Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SPONDYLARTHRITIS COHORT
  Interventions: Other: Imaging exams

INTERVENTIONS:
Other: Imaging exams — Radiological examinations:
  * Standard x-ray: they include an x-ray of the cervical, thoracic, and lumbar spine (side-on), of the lumbar spine from the front and an x-ray of the pelvis from the front
  * MRI scan: are taken of the cervical, thoracic and lumbar spine and sacroiliac joints.
  Bone densitometry: evaluation of bone densitometry of the lumbar spine and femoral neck.
  Enthesis ultrasound: bilateral evaluation of entheseal insertions for the Achilles tendon, patella tendons and epicondyle tendons.
  Biological tests :
  * Genetic test : DNA will be collected at the first visit from all centers. RNA will be collected at the inclusion visit in AP-HP centres only.
  * Serum will be collected by all centres at the initial visit, then in M6, M12 and M24 for the first two years of the study, then in M60.
  * Urine will be collected by all centres at the initial visit, then in M24 for the first two years of the study, then in M60.
  Other Names: Radiological examinations; Bone densitometry; Enthesis ultrasound; Biological tests

SUMMARY:
This study is a large national multicenter, longitudinal, prospective follow-up of patients presenting with early inflammatory back pain in order to set up a database to facilitate several investigations on diagnosis, prognosis, epidemiology, pathogenesis and medico-economics in the field of early inflammatory back pain and spondyloarthritis

DETAILED DESCRIPTION:
This large national multicenter, longitudinal, prospective follow-up of patients presenting with early inflammatory back pain in order to set up a database to facilitate several investigations on diagnosis, prognosis, epidemiology, pathogenesis and medico-economics in the field of early inflammatory back pain and spondyloarthritis.

The Patients were recruited if they had inflammatory back pain of more than 3months and less than 3years. Patients will be followed every 6months during the first 2years then every year during at least 5years. Apart from information collected on a Case Report Form (demographics, disease activity, severity, co-morbidities, socio-economics, treatments, radiological and MRI evaluation of the spine and the pelvis according to the local investigators, and for some centers bone densitometry and ultrasonography of entheses), the digital X-rays and MRI of the spine and pelvis are stored using a specific software (Carestream) and the biological samples (DNA, RNA, sera, urines) are centralized at the Biological Resources Center (Bichat Hospital).

This large cohort should facilitate the conduct of researches in different areas (clinical, medico-economics, translational) in order to improve our knowledge on the pathogenesis and natural history of axial spondyloarthritis

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 and under 50 years
* Inflammatory back pain (buttock, lumbar or thoracic spine) fulfilling either the Calin orBerlin criteria :
* Calin criteria (at least 4 of 5 criteria must be met) (ref. 25):
* Insidious onset
* Onset before age 40
* Persistence since at least three months
* Morning stiffness 30 minutes
* Improvement with exercise
* Berlin criteria (at least 2 of 4 criteria must be met) (ref. 26):
* Morning stiffness 30 minutes
* Improvement with exercise and absence of improvement at rest
* Nocturnal pain in the second part of the night
* Alternating buttock pain
* Symptom duration more than 3 months and less than 3 years
* Symptoms suggestive of spondyloarthritis according to the local investigator's assessment(e.g. score ≥5 on a 0 to 10 numerical rating scale in which 0 = no suggestive and 10 = verysuggestive of spondyloarthritis)
* Realization of a prior medical examination (article L.1121-11 of the Code of the Public health)
* Informed consent Dated and signed voluntarily

Exclusion Criteria:

* Other spinal disease clearly defined (eg symptomatic mechanical discopathy)
* Pregnant woman
* History of alcoholism, drug addiction, psychological problems, severe co-morbidities which might interfere with the validity of the informed consent and/or prevent an optimal compliance of the patient to the cohort
* It was possible to include patients who have received or are receiving a thorough treatment such as Sulfasalazine, Methotrexate or Azathioprine. However any history of treatment with biotherapy including anti-TNF therapy defined exclusion criteria
* Corticosteroid intake was permitted only in case of a dose lower than 10 mg prednisoneper day and stable for at least 4 weeks prior baseline
* MRI contraindication
* No affiliation to the French National Social Security System

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients presenting early inflammatory back pain of more than 3 months and less than 3 years
Sampling Method: Non-Probability Sample
Enrollment: 708 (Actual)
Dates: Start 2007-10-15 (Actual); Primary Completion 2016-06-20 (Actual); Study Completion 2022-02-23 (Actual)

PRIMARY OUTCOMES:
Radiological sacroiliitis | 5 years
  Percentage of patients after 5 years of evolution, that will have a radiological sacroiliitis according to the presence or absence of the sacroiliac inflammatory abnormalities of the sacroiliac joints at study entry on MRI

SECONDARY OUTCOMES:
Predictive biomarker(s) of structural radiographic or IRM progression in SpA | 5 years
  To identify biomarker(s) of bone formation (DKK-1, sclérostin, BMP-7, périostin) which are predictive of structural radiographic progression and in IRM at 5 years
Changes of level of biomarkers in the disease in 5 years | 5 years
  To assess the 5-year changes in of serum periostin, serum sclerostin, DKK-1 and BMP-7 in a large population of early axial SpA
Changes of level of biomarkers in the disease in 2 years | 2 years
  To assess the 2-year changes in of serum periostin, serum sclerostin, DKK-1 and BMP-7 in a large population of early axial SpA
Correlation and/or association between changes of biomarkers and structural damages at 2 and 5 years | 5 years
Correlation and/or association between changes of biomarkers and disease activity at 2 and 5 years | 5 years
Correlation and/or association between changes of biomarkers in patients with or without anti-TNF treatment | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Maxime DOUGADOS, MD, Principal Investigator — Cochin Hospital
Locations (1):
- Department of Rheumatology, Cochin Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dougados M, d'Agostino MA, Benessiano J, Berenbaum F, Breban M, Claudepierre P, Combe B, Dargent-Molina P, Daures JP, Fautrel B, Feydy A, Goupille P, Leblanc V, Logeart I, Pham T, Richette P, Roux C, Rudwaleit M, Saraux A, Treluyer JM, van der Heijde D, Wendling D. The DESIR cohort: a 10-year follow-up of early inflammatory back pain in France: study design and baseline characteristics of the 708 recruited patients. Joint Bone Spine. 2011 Dec;78(6):598-603. doi: 10.1016/j.jbspin.2011.01.013. Epub 2011 Mar 31. PMID 21458351
- [Derived] Maksymowych WP, Claudepierre P, de Hooge M, Lambert RG, Landewe R, Molto A, van der Heijde D, Bukowski JF, Jones H, Pedersen R, Szumski A, Vlahos B, Dougados M. Erosions on T1-Weighted Magnetic Resonance Imaging Versus Radiography of Sacroiliac Joints in Recent-Onset Axial Spondyloarthritis: 2-Year Data (EMBARK Trial and DESIR Cohort). J Rheumatol. 2024 May 1;51(5):462-471. doi: 10.3899/jrheum.2023-0906. PMID 38359938
- [Derived] Aouad K, Tournadre A, Lucasson F, Wendling D, Molto A, Fautrel B, Gossec L. Influence of Sex on Early Axial Spondyloarthritis: A Six-Year Longitudinal Analysis From a Large National Cohort. Arthritis Care Res (Hoboken). 2023 Oct;75(10):2107-2116. doi: 10.1002/acr.25103. Epub 2023 Mar 15. PMID 36785996
- [Derived] Ruyssen-Witrand A, Rousseau V, Sommet A, Goupille P, Degboe Y, Constantin A. Factors associated with drug-free remission at 5-year in early onset axial spondyloarthritis patients: Data from the DESIR cohort. Joint Bone Spine. 2022 Jul;89(4):105358. doi: 10.1016/j.jbspin.2022.105358. Epub 2022 Feb 12. PMID 35167972
- [Derived] Lucasson F, Richette P, Aouad K, Ryussen-Witrand A, Wendling D, Fautrel B, Gossec L. Prevalence and consequences of psoriasis in recent axial spondyloarthritis: an analysis of the DESIR cohort over 6 years. RMD Open. 2022 Jan;8(1):e001986. doi: 10.1136/rmdopen-2021-001986. PMID 35091462
- [Derived] Costantino F, Aegerter P, Schett G, De Craemer AS, Molto A, Van den Bosch F, Elewaut D, Breban M, D'Agostino MA. Cluster analysis in early axial spondyloarthritis predicts poor outcome in the presence of peripheral articular manifestations. Rheumatology (Oxford). 2022 Aug 3;61(8):3289-3298. doi: 10.1093/rheumatology/keab873. PMID 34864930
- [Derived] Kumaradev S, Roux C, Sellam J, Perrot S, Pham T, Dugravot A, Molto A. Socio-demographic determinants in the evolution of pain in inflammatory rheumatic diseases: results from ESPOIR and DESIR cohorts. Rheumatology (Oxford). 2022 Apr 11;61(4):1496-1509. doi: 10.1093/rheumatology/keab562. PMID 34270700
- [Derived] Maksymowych WP, Claudepierre P, de Hooge M, Lambert RG, Landewe R, Molto A, van der Heijde D, Bukowski JF, Jones H, Pedersen R, Szumski A, Vlahos B, Dougados M. Structural changes in the sacroiliac joint on MRI and relationship to ASDAS inactive disease in axial spondyloarthritis: a 2-year study comparing treatment with etanercept in EMBARK to a contemporary control cohort in DESIR. Arthritis Res Ther. 2021 Jan 29;23(1):43. doi: 10.1186/s13075-021-02428-8. PMID 33514428
- [Derived] Carvalho PD, Ruyssen-Witrand A, Marreiros A, Machado PM. Long-Term Association Between Disease Activity and Disability in Early Axial Spondyloarthritis: Results From a Prospective Observational Study of Inflammatory Back Pain. Arthritis Care Res (Hoboken). 2022 May;74(5):768-775. doi: 10.1002/acr.24515. Epub 2022 Mar 7. PMID 33207078
- [Derived] Descamps E, Molto A, Borderie D, Lories R, Richard CM, Pons M, Roux C, Briot K. Changes in bone formation regulator biomarkers in early axial spondyloarthritis. Rheumatology (Oxford). 2021 Mar 2;60(3):1185-1194. doi: 10.1093/rheumatology/keaa296. PMID 32888036
- [Derived] Lopez-Medina C, Molto A, Claudepierre P, Dougados M. Clinical manifestations, disease activity and disease burden of radiographic versus non-radiographic axial spondyloarthritis over 5 years of follow-up in the DESIR cohort. Ann Rheum Dis. 2020 Feb;79(2):209-216. doi: 10.1136/annrheumdis-2019-216218. Epub 2019 Nov 29. PMID 31784451
- [Derived] Ruyssen-Witrand A, Luxembourger C, Cantagrel A, Nigon D, Claudepierre P, Degboe Y, Constantin A. Association between IL23R and ERAP1 polymorphisms and sacroiliac or spinal MRI inflammation in spondyloarthritis: DESIR cohort data. Arthritis Res Ther. 2019 Jan 15;21(1):22. doi: 10.1186/s13075-018-1807-5. PMID 30646942
- [Derived] Dougados M, Maksymowych WP, Landewe RBM, Molto A, Claudepierre P, de Hooge M, Lambert RG, Bonin R, Bukowski JF, Jones HE, Logeart I, Pedersen R, Szumski A, Vlahos B, van der Heijde D. Evaluation of the change in structural radiographic sacroiliac joint damage after 2 years of etanercept therapy (EMBARK trial) in comparison to a contemporary control cohort (DESIR cohort) in recent onset axial spondyloarthritis. Ann Rheum Dis. 2018 Feb;77(2):221-227. doi: 10.1136/annrheumdis-2017-212008. Epub 2017 Sep 29. PMID 28970213
- [Derived] Ruyssen-Witrand A, Jamard B, Cantagrel A, Nigon D, Loeuille D, Degboe Y, Constantin A. Relationships between ultrasound enthesitis, disease activity and axial radiographic structural changes in patients with early spondyloarthritis: data from DESIR cohort. RMD Open. 2017 Sep 7;3(2):e000482. doi: 10.1136/rmdopen-2017-000482. eCollection 2017. PMID 28955496
- [Derived] Ez-Zaitouni Z, Hilkens A, Gossec L, Berg IJ, Landewe R, Ramonda R, Dougados M, van der Heijde D, van Gaalen F. Is the current ASAS expert definition of a positive family history useful in identifying axial spondyloarthritis? Results from the SPACE and DESIR cohorts. Arthritis Res Ther. 2017 May 31;19(1):118. doi: 10.1186/s13075-017-1335-8. PMID 28569222
- [Derived] Molto A, Tezenas du Montcel S, Wendling D, Dougados M, Vanier A, Gossec L. Disease activity trajectories in early axial spondyloarthritis: results from the DESIR cohort. Ann Rheum Dis. 2017 Jun;76(6):1036-1041. doi: 10.1136/annrheumdis-2016-209785. Epub 2016 Nov 25. PMID 27888172
- [Derived] Canoui-Poitrine F, Poulain C, Molto A, Le Thuaut A, Lafon C, Farrenq V, Ferkal S, Le Corvoisier P, Ghaleh B, Bastuji-Garin S, Fautrel B, Dougados M, Claudepierre P. Early tumor necrosis factor alpha antagonist therapy in everyday practice for inflammatory back pain suggesting axial spondyloarthritis: results from a prospective multicenter french cohort. Arthritis Care Res (Hoboken). 2014 Sep;66(9):1395-402. doi: 10.1002/acr.22330. PMID 24664935